CLINICAL TRIAL: NCT06576089
Title: Optimizing Recruitment to Drive Equitable Research Opportunity in Stroke Rehabilitation in Canada - The ORDER Pilot Study
Brief Title: Optimizing Recruitment to Drive Equitable Research Opportunity in Stroke Rehabilitation Trials in Canada
Acronym: ORDER-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ada Tang, Professor, Assistant Dean, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ORDER-Pilot
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; Clinical trial; Informed consent; Diversity, Equity, Inclusion; Sex
MeSH Terms: conditions — Stroke; Coitus | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional recruitment and enrollment processes (TRAD) (Other): Traditional participant information letter and consent form only (TRAD)
  Interventions: Other: Traditional recruitment and enrollment processes (TRAD)
- Supported, women-centred and aphasia-friendly recruitment and enrollment process (ORDER) (Experimental): Supplementing traditional recruitment methods (detailed participant information letter and consent form) with women-centred, aphasia-friendly recruitment video and leaflet (ORDER)
  Interventions: Other: Supported, women-centred and aphasia-friendly recruitment and enrollment process (ORDER)

INTERVENTIONS:
Other: Supported, women-centred and aphasia-friendly recruitment and enrollment process (ORDER) — Participants randomized into ORDER will be approached by the Site Coordinator for interest in the host trial. The Coordinator will introduce the trial and share a brief, women-centred, aphasia-friendly, close-captioned video that further describes the trial procedures and an accompanying leaflet.
  ORDER recruitment materials will be saved to a mobile tablet. The Coordinator will watch the video together with the potential participant, engage in discussion about the host trial and answer any questions they may have. The Coordinator will offer to leave the tablet with the potential participant, along with printed copies of the leaflet and participant information letter. The Coordinator will encourage them to share these materials with their family members, friends or member of their healthcare team who may assist with decision making. The Coordinator will return in the following days to address any further questions and determine the decision whether to enroll in the trial.
  Arms: Supported, women-centred and aphasia-friendly recruitment and enrollment process (ORDER)
Other: Traditional recruitment and enrollment processes (TRAD) — Participants randomized into the traditional recruitment process (TRAD) will be approached by the Site Coordinator for interest in the CAMAROS trial and presented with the standard participant information letter and full informed consent form. The information letter and consent form will be left with the potential participant to view again; the Coordinator will encourage them to share these materials with their family members or friends who may assist with decision making. The Coordinator will return in the following days to address any further questions and determine the decision whether to enroll in the trial.
  Arms: Traditional recruitment and enrollment processes (TRAD)

SUMMARY:
Stroke is a major health issue in Canada. Stroke affects over 400,000 Canadians, and this number is expected to nearly double by 2038. Research studies in stroke recovery can help us better understand effective rehabilitation treatments and help reduce the burden of stroke. Some groups of people however are commonly not included in stroke studies. For example, it is more common for men to take part in research than women, and people with aphasia (a language impairment commonly seen after stroke) are often excluded from studies. Also, deciding whether to even take part in a research study can be difficult and overwhelming, especially in the early days after stroke, leaving many people to decline to participate. Research has shown that women experience different barriers to participating in stroke research than men. This means that research findings, and the decisions made during stroke care based on these findings, may not reflect the true stroke population. Better ways to help support groups like women and people with aphasia to participate in stroke research are needed, so that study findings will better represent people living with stroke.

DETAILED DESCRIPTION:
Clinical trials in stroke recovery are essential for establishing effective treatments, yet important groups, such as women and people with aphasia, have been consistently under-represented in stroke trials. This limits the generalizability of trial findings and impacts clinical care. Relevant to stroke is the critical time window for neuroplastic change that makes timely enrolment into stroke recovery trials of particular importance. There is a need to develop strategies to efficiently and effectively promote participation into stroke recovery trials.

The Optimizing Recruitment to Drive Equitable Research opportunity in stroke rehabilitation trials in Canada (ORDER) is a pilot "study within a trial" to look at a women-centred, aphasia-friendly recruitment method for a research trial examining whether a medication (Maraviroc), when combined with rehabilitation, can help with stroke recovery ("host trial").

The objectives of this pilot study are to:

1. Examine the feasibility of a women-centred, aphasia-friendly video and leaflet (ORDER) to supplement traditional detailed participant information letters, support recruitment, and drive enrollment in a stroke recovery randomized trial;
2. Understand the barriers and facilitators associated with enrolling in the host trial and stroke recovery trials more broadly;
3. Determine preliminary estimates of effect of ORDER compared to traditional recruitment and enrollment processes

The study will take place at the 10 sites across 6 provinces. The host trial is comparing Maraviroc vs. placebo, combined with 8 weeks of rehabilitation, to improve motor and sensory function.

Potential participants will be identified and approached 5 days to 8 weeks after stroke and randomized to: 1) Supplementing traditional recruitment methods (detailed participant information letter and consent form) with women-centred, aphasia-friendly recruitment video and leaflet (ORDER), or 2) Traditional participant information letter and consent form only (TRAD). For the ORDER arm, the video and leaflet will be saved to a tablet and reviewed together with the Coordinator and potential participant. The Coordinator will engage in discussion about the host trial (prompting questions will be provided), and will offer to leave the tablet with the person, along with printed copies of the leaflet and participant information letter. They will be encouraged to share these materials with their family members or friends who may assist with decision making. For TRAD, the Coordinator will review the information letter and consent form, offer to leave these with the person to view again, and encourage them to share these materials with their family members or friends who may assist with decision making. For both arms, the Coordinator will return in the following days to address any further questions and determine the decision whether to enroll in the trial.

Objective 1 Feasibility will be determined as enrollment (# consented/approached, # women consented/total # consented) and efficiency (# days to decision, # interactions between Site Coordinator and potential participants), with a priori criteria for success for each indicator.

For Objective 2 (Barriers and facilitators), individuals will be invited to complete a survey or participate in key-informant, semi-structured interviews (15 enrolled, 15 declined, 10 Site Coordinators) to share their perceptions of the enrollment and consent process, reason(s) for declining to participate, and recruitment reach (# and characteristics of individuals enrolled through ORDER and TRAD). Purposive sampling will be used to obtain diversity across sex (males, females), gender (men, women, transgender, non-binary), and racial background and will train peer researchers with lived experience to conduct the interviews. The interview guide will be co-developed with our patient partners and the research team. Deductive content analysis of interview transcripts will be conducted and mapped to the Theoretical Domains Framework.

For Objective 3 (Preliminary estimates of effect), enrollment and efficiency will be compared between ORDER and TRAD, and Cohen's d and f will be calculated for unadjusted and adjusted analyses to help inform future large-scaled trials.

ELIGIBILITY:
Inclusion Criteria:

1. Primary ischemic anterior circulation stroke
2. Age ≥18 years
3. ≥5 days but <8 weeks after stroke on the date of medication (Maraviroc or placebo) start
4. Hemiparesis requiring inpatient rehabilitation
5. Assistance available for daily rehabilitation training practice and for transportation when needed
6. Adequate language skills to understand Informed Consent and retain information during daily therapies
7. At least one of the following: some shoulder abduction with gravity eliminated and visible extension in two or more digits OR visible hip flexion or extension

Exclusion Criteria:

1. Pre-stroke modified Rankin score ≥2
2. Limited resources or illness that will not enable a return to living outside of a facility
3. History of dementia
4. History of hepatitis or elevated hepatic transaminases or bilirubin
5. History of renal insufficiency or creatinine clearance (eGFR) <60mL / min / 1.73m2
6. Cancer or other chronic illness that makes 1-year survival unlikely or will detract from the ability to carry out exercise and skills practice
7. Existing pre-stroke serious disabling disease (e.g., Parkinson's disease, severe traumatic brain injury, amputation)
8. Seizure related to stroke
9. Acute or chronic epilepsy
10. Currently taking any of the following anticonvulsant medications: Carbamazepine, Phenobarbital, Phenytoin
11. Pregnant, breastfeeding, or positive test for pregnancy at baseline
12. Women of childbearing potential who are not using one highly effective form of contraception or two forms of effective contraception
13. Known HIV positivity
14. Currently taking any of the following antifungal and/or antibacterial medications: Ketoconazole, Itraconazole, Voriconazole, Rifampin, Clarithromycin, Rifabutin + Protease Inhibitor
15. Currently taking St. John's Wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From date identified as eligible for the host trial to date of decision (consent or decline)
  Each site will record # patients approached, # consented (by men and women), date of initial contact by the Site Coordinator, date of decision (consent or decline), and # interactions between the Site Coordinator and potential participants for ORDER and TRAD.
Barriers and facilitators | From date of decision (consent or decline) for host trial to date of survey or interview
  Short survey and semi-structured interviews to examine the perceptions of the enrollment and consent process of individuals approached to participate in CAMAROS and Site Coordinators. Reason(s) for declining to participate and recruitment reach (# and characteristics of individuals approached for CAMAROS) will also be recorded.
Preliminary estimates of effect | From date identified as eligible for the host trial to date of decision (consent or decline)
  Each site will record # patients approached, # consented (by men and women), date of initial contact by the Site Coordinator, date of decision (consent or decline), and # interactions between the Site Coordinator and potential participants for ORDER and TRAD.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - University of Calgary & Foothills Medical Centre, Calgary, Alberta
  - University of British Columbia & GF Strong Rehabilitation Centre, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - Parkwood Institute, London, Ontario
  - Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario